CLINICAL TRIAL: NCT00844792
Title: A Randomized, Double-Blind Study of Combination Vitamin E, Selenium and Lycopene vs. Placebo in Men Undergoing Radical Prostatectomy for Prostate Cancer
Brief Title: Study of Antioxidants on Prostate Tumors in Men Undergoing Radical Prostatectomy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-0604-CE
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cancer of the Prostate; Prostate Cancer; Prostatic Neoplasms
Keywords: Male Urogenital Diseases; Antioxidants; Vitamin E; Vitamin D; Lycopene; Selenium
MeSH Terms: conditions — Prostatic Neoplasms; Male Urogenital Diseases | interventions — Lycopene; Cholecalciferol; Selenium; Tea; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This group of men will be on active treatment (antioxidants)for 6-8 weeks prior to their radical prostatectomy.
  Interventions: Dietary Supplement: Lycopene, Vitamin D3, Selenium, Green Tea Extract, Vitamin E
- 2 (Placebo Comparator): This group of men will be on placebo for 6-8 weeks prior to their radical prostatectomy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Lycopene, Vitamin D3, Selenium, Green Tea Extract, Vitamin E — Twice a day with meals. Lycopene - 20 mg, Vitamin D3 - 200 IU, Selenium - 100 mcg, Green Tea Extract - 75 mg, Vitamin E - 50 IU
  Arms: 1
Drug: Placebo — Twice a day with meals.
  Arms: 2

SUMMARY:
The purpose of this study is to see if an intervention of antioxidants(vitamin E, selenium and lycopene) can change (reduce) prostate tumor size and alter certain markers that can affect tumor growth and prostate cancer aggressiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Gleason score > or = to 7 adenocarcinoma of the prostate
* At least 30% of one core involved
* Radical prostatectomy planned
* Willingness to discontinue use of supplements at least 4 weeks prior to study intervention (for subjects using vitamin E, selenium or lycopene at time of consent)
* ability and willingness to consume study intervention for 6 - 8 weeks prior to radical prostatectomy.

Exclusion Criteria:

* Previous treatment for prostate cancer
* Current use of finasteride or dutasteride

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the impact of combination Vitamin E, Selenium and Lycopene on prostate tumor size and to study certain markers in blood and prostate tissue which affect prostate tumor growth or shrinkage. | Blood samples will be collected prior to intervention and 8 weeks later , prior to surgery. Prostate tissue will be harvested at time of surgery, after the prostate has been removed.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada